CLINICAL TRIAL: NCT03682107
Title: A Phase I, Randomized, Placebo Controlled, Double-Blind, Dose Escalation Trial to Evaluate the Safety and Immunogenicity of an Andes Virus DNA Vaccine for the Prevention of Hantavirus Pulmonary Syndrome Using the PharmaJet Stratis(R) Needle-Free Injection System in Normal Healthy Adults
Brief Title: Andes Virus DNA Vaccine for the Prevention of Hantavirus Pulmonary Syndrome Using the PharmaJet Stratis(R) Needle-Free Injection Delivery Device
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16-0119; HHSN272201300016I
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Results first posted 2021-10-14 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2021-04-06

CONDITIONS: Hantavirus Pulmonary Infection; Immunisation
Keywords: Andes Virus DNA; ANDV DNA; Hantavirus; Immunogenicity; PharmaJet Stratis; Pulmonary Syndrome; Safety; Vaccine
MeSH Terms: conditions — Hantavirus Pulmonary Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1 (2 mg ANDV - 3-dose regimen) (Experimental): 1 sentinel subject assigned to the 3-dose regimen will receive 2 mg (2 injections of 0.5 ml (1 mg/0.5 ml each)) of ANDV DNA vaccine intramuscularly into the left and right deltoid on Day 1 in an open label manner, and 2 mg (2 injections of 0.5 ml (1 mg/0.5 ml each)) of ANDV DNA vaccine on Days 29, 169, and matching placebo on Day 57 in double-blind manner.
  11 subjects assigned to the 3-dose regimen will receive either 2 mg (2 injections of 0.5 ml (1 mg/0.5 ml each)) of ANDV DNA vaccine intramuscularly into the left and right deltoid on Days 1, 29, 169, and matching placebo on Day 57 (n=9) or matching placebo on Days 1, 29, 57, and 169 (n=2).
  Interventions: Biological: Andes virus DNA vaccine; Other: Placebo
- Arm 2 (2 mg ANDV - 4-dose regimen) (Experimental): 1 sentinel subject assigned to the 4-dose regimen will receive 2 mg (2 injections of 0.5 ml (1 mg/0.5 ml each)) of ANDV DNA vaccine intramuscularly into the left and right deltoid on Day 1 in an open label manner, and Days 29, 57 and 169 in double-blind manner.
  11 subjects assigned to the 4-dose regimen will receive either 2 mg (2 injections of 0.5 ml (1 mg/0.5 ml each)) of ANDV DNA vaccine intramuscularly into the left and right deltoid on Days 1, 29, 57 and 169 (n=9) or matching placebo on Days 1, 29, 57, and 169 (n=2).
  Interventions: Biological: Andes virus DNA vaccine; Other: Placebo
- Arm 3 (4 mg ANDV - 3-dose regimen) (Experimental): 1 sentinel subject assigned to the 3-dose regimen will receive 4 mg (2 injections of 0.5 ml (2 mg/0.5 ml each)) of ANDV DNA vaccine intramuscularly into the left and right deltoid on Day 1 in an open label manner, and 4 mg (2 injections of 0.5 ml (2 mg/0.5 ml each)) of ANDV DNA vaccine on Days 29, 169, and matching placebo on Day 57 in double-blind manner.
  11 subjects assigned to the 3-dose regimen will receive either 4 mg (2 injections of 0.5 ml (2 mg/0.5 ml each)) of ANDV DNA vaccine intramuscularly into the left and right deltoid on Days 1, 29, 169, and matching placebo on Day 57 (n=9) or matching placebo on Days 1, 29, 57, and 169 (n=2).
  Interventions: Biological: Andes virus DNA vaccine; Other: Placebo
- Arm 4 (4 mg ANDV - 4-dose regimen) (Experimental): 1 sentinel subject assigned to the 4-dose regimen will receive 4 mg (2 injections of 0.5 ml (2 mg/0.5 ml each)) of ANDV DNA vaccine intramuscularly into the left and right deltoid on Day 1 in an open label manner, and Days 29, 57 and 169 in double-blind manner.
  11 subjects assigned to the 4-dose regimen will receive either 4 mg (2 injections of 0.5 ml (2 mg/0.5 ml each)) of ANDV DNA vaccine intramuscularly into the left and right deltoid on Days 1, 29, 57 and 169 (n=9) or matching placebo on Days 1, 29, 57, and 169 (n=2).
  Interventions: Biological: Andes virus DNA vaccine; Other: Placebo

INTERVENTIONS:
Biological: Andes virus DNA vaccine — A vaccine targeting the hantavirus pulmonary syndrome (HPS) causative agent Andes Virus (ANDV), with potential pan-hantavirus effect. The plasmid backbone, pWRG7077, is modified to produce the active ingredient of the vaccine, plasmid pWRG/AND-M (opt2), and includes the ANDV M gene responsible for encoding viral GnGc envelope glycoproteins. ANDV DNA vaccine will be administered intramuscularly at 2 mg or 4 mg doses using the PharmaJet Stratis Needle-Free Injection System.
Other: Placebo — Normal saline injections will be administered intramuscularly as matching placebo using the PharmaJet Stratis Needle-Free Injection System

SUMMARY:
This is a Phase 1, randomized, placebo controlled, double-blind, dose escalation trial of 48 males and non-pregnant females, 18-49 years old, inclusive, who are in good health and meet all eligibility criteria. This trial is designed to assess the safety, reactogenicity and immunogenicity of an Andes Virus (ANDV) DNA vaccine for the prevention of Hantavirus Pulmonary Syndrome (HPS). ANDV DNA vaccine or placebo will be administered using the PharmaJet Stratis(R) Needle-Free Injection System. The study duration is 23 months while the subject participation duration is 12 months. Subjects assigned to the 3 dose regimen will receive ANDV DNA vaccine on Days 1, 29 and 169, and placebo on Day 57. Subjects assigned to the 4 dose regimen will receive ANDV DNA on Days 1, 29, 57 and 169. Two doses (2 or 4 mg) of ANDV DNA vaccine will be evaluated. The primary objective of this study is to assess the safety and reactogenicity of the ANDV DNA vaccine by dosage cohort and treatment arm when administered using the PharmaJet Stratis(R) Needle-Free Injection system in normal, healthy adults.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, placebo controlled, double-blind, dose escalation trial of 48 males and non-pregnant females, 18-49 years old, inclusive, who are in good health and meet all eligibility criteria. This trial is designed to assess the safety, reactogenicity and immunogenicity of an Andes Virus (ANDV) DNA vaccine for the prevention of Hantavirus Pulmonary Syndrome (HPS). ANDV DNA vaccine or placebo will be administered using the PharmaJet Stratis(R) Needle-Free Injection System. The study duration is 23 months while the subject participation duration is 12 months. Subjects assigned to the 3 dose regimen will receive ANDV DNA vaccine on Days 1, 29 and 169, and placebo on Day 57. Subjects assigned to the 4 dose regimen will receive ANDV DNA on Days 1, 29, 57 and 169. Two doses (2 or 4 mg) of ANDV DNA vaccine will be evaluated. The primary objective of this study is to assess the safety and reactogenicity of the ANDV DNA vaccine by dosage cohort and treatment arm when administered using the PharmaJet Stratis(R) Needle-Free Injection system in normal, healthy adults. The secondary objective of this study is to assess the immunogenicity of the ANDV DNA vaccine by dosage cohort and treatment arm.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent before initiation of any study procedures.
2. Are able to understand and comply with planned study procedures and be available for all study visits/phone calls.
3. Males or non-pregnant females ages 18-49, inclusive.
4. Are in good health*. *As determined by medical history and physical examination to evaluate acute or currently ongoing chronic medical diagnoses or conditions, defined as those that have been present for at least 90 days which would affect the assessment of the safety of subjects or the immunogenicity of study vaccinations. Chronic medical diagnoses or conditions should be stable for the last 60 days (no hospitalizations, ER or urgent care for condition and no adverse symptoms that need medical intervention such as medication change/supplemental oxygen). This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis or condition in the 60 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening of medical diagnosis or condition. Similarly, medication changes subsequent to enrollment and study vaccination are acceptable provided there was no deterioration in the subject's chronic medical condition that necessitated a medication change, and there is no additional risk to the subject or interference with the evaluation of responses to study vaccination. Note: Topical, nasal, and inhaled medications (apart from steroids as outlined in the Subject Exclusion Criteria), herbals, vitamins, and supplements are permitted.
5. Oral temperature is less than 100.0 degrees Fahrenheit (37.8 degrees Celsius).
6. Pulse is 47 to 105 beats per minute (bpm), inclusive.
7. Systolic blood pressure (BP) is 85 to 150 mm Hg, inclusive.
8. Diastolic blood pressure (BP) is 55 to 95 mm Hg, inclusive.
9. Have acceptable screening laboratories* within 28 days prior to enrollment. *Screening laboratory values that are outside acceptable range but are thought to be due to an acute condition or due to laboratory error may be repeated once.
10. Urine protein screen is negative or trace.
11. Drug screen for opiates is negative.
12. HgbA1C < 6.3% at screening.
13. HIV - 1/2 antibody negative.
14. HCV antibody negative.
15. HBsAg negative.
16. Women of childbearing potential*, must be using an effective method of contraception** from 30 days prior to the first study vaccination until 90 days after the last study vaccination.

    *Women of childbearing potential are defined as those who have not been sterilized via tubal ligation, bilateral oophorectomy, hysterectomy, or successful Essure(R) placement (permanent, non-surgical, non-hormonal sterilization) with history of documented radiological confirmation test at least 90 days after the procedure (or with use of another birth control method if history of confirmation test not confirmed), AND are still menstruating or < 1 year since the last menses if perimenoapausal.

    **For this study, we define an effective contraceptive method as one that results in a failure rate of less than 1% per year when it is used consistently and correctly. This includes, but is not limited to, non-male sexual relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with a vasectomized partner, male condoms with the use of applied spermicide, intrauterine devices, NuvaRing(R), and licensed hormonal methods such as implants, injectables or oral contraceptives ("the pill").
17. Women of childbearing potential* must have a negative serum pregnancy test at screening and a negative urine pregnancy test within 24 hours prior to each study vaccination.

    *See definition of women of childbearing potential above.
18. Sexually active male participants whose partner is a woman of childbearing potential* and has not had a vasectomy** must agree not to father a child until 90 days after the last vaccination***.

    * See definition of women of childbearing potential above. **Performed > 1 year prior to screening

      * Must agree to use a barrier method of birth control e.g., either condom with spermicidal foam/gel/film/cream or partner reports usage of occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
19. Women agree to not donate eggs (ova, oocytes) and male subject agrees not to donate sperm from the start of screening onwards until at least 90 days after the last vaccination.
20. Agree not to participate in another clinical trial during the study period.
21. Agree not to donate blood to a blood bank for 3 months after receiving the last study vaccine.

Exclusion Criteria:

1. Women who are pregnant, planning to become pregnant or lactating*. *Includes breastfeeding or planning to breastfeed at any given time from the receipt of study vaccination through the 12-month trial period.
2. Known allergy or history of anaphylaxis, severe local or other serious adverse reactions to vaccines or vaccine products*, or history of severe allergic reactions.

   *This includes a known allergy to an aminoglycoside (e.g., gentamicin, tobramycin, neomycin, streptomycin).
3. Received an experimental agent* within 3 months prior to study vaccination, or expects to receive an experimental agent** during the 12-month trial-reporting period.

   *Including vaccine, drug, biologic, device, blood product, or medication.

   **Other than from participation in this study.
4. Received any licensed live vaccine within 28 days prior to or after each study vaccination.
5. Received a licensed inactivated vaccine within 14 days prior to or after each study vaccination*.

   *Allowable exception for inactivated seasonal influenza vaccine received more than 7 days prior to or after a study vaccination.
6. Individuals in whom the ability to observe possible local reactions at the eligible injection sites (deltoid region) is, unacceptably obscured due to a physical condition or permanent body art.
7. Have an acute illness*, as determined by the site PI or appropriate sub-investigator, within 72 hours prior to study vaccination.

   *An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol. Subjects may re-screen after an acute illness is resolved
8. Any confirmed or suspected immunosuppressive or immunodeficient condition* or use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.

   *Including HIV infection
9. Administration of chronic (defined as more than 14 days) immunosuppressants or other immune modifying drugs within 6 months of receipt of study vaccine*.

   *For corticosteroids, this means prednisone, or equivalent, greater than or equal to 0.5 mg/kg/day. Intranasal and topical steroids ARE allowed; daily inhaled steroids for treatment of asthma NOT allowed.
10. History of receipt of a Hantavirus vaccine, including vaccines for Hantaan virus, Puumala virus, or combination of both.
11. Exposed to ANDV* or plans to travel to an endemic area** from enrollment through 6 months post last vaccination.

    *Residence in an ANDV endemic area in the last 3 years or > 2 consecutive weeks of travel to an ANDV endemic area** in the last 3 years.

    **ANDV endemic areas include Chile, Brazil and Argentina.
12. Any chronic or active neurologic disorder, including seizures and epilepsy, excluding febrile seizures as a child.
13. History of receiving immunoglobulin or other blood product within the 3 months before enrollment in this study.
14. Current or past history of alcohol or drug abuse in the last 5 years.
15. Subjects with autoimmune disorders, chronic inflammatory disorders or neurological disorders with a potential autoimmune correlation.
16. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.
17. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 10 years prior to study vaccination.
18. Have received any antiviral within 3 days of study vaccination.
19. A diagnosis of Type I or II diabetes.
20. Current employee or staff paid entirely or partially by the contract for this trial, or staff who are supervised by the PI or Sub-Investigators.
21. Any condition that would, in the opinion of the Site Investigator or appropriate sub-investigator, is a contraindication to study participation*.

    * Including acute or chronic (persisting for at least 90 days) clinically significant medical disease or condition, that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of the study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Paulsen GC, Frenck R Jr, Tomashek KM, Alarcon RM, Hensel E, Lowe A, Brocato RL, Kwilas SA, Josleyn MD, Hooper JW. Safety and Immunogenicity of an Andes Virus DNA Vaccine by Needle-Free Injection: A Randomized, Controlled Phase 1 Study. J Infect Dis. 2024 Jan 12;229(1):30-38. doi: 10.1093/infdis/jiad235. PMID 37380156

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population includes 48 males and non-pregnant females, 18-49 years old, inclusive, who are in good health, have not previously received the Hantavirus vaccine, have not been exposed to ANDV, and meet all other eligibility criteria. Participants were enrolled between 19FEB2019 and 04NOV2019 and received study vaccinations between 19FEB2019 and 08APR2020.
Groups:
- 2 mg ANDV, 3 Dose Regimen: 2 mg (2 injections of 0.5 mL (1 mg/0.5 mL each)) of ANDV DNA vaccine intramuscularly into the left and right deltoid on Days 1, 29, and 169 in a double-blinded manner. Sentinel subjects received all doses in an open label manner.
  Andes virus DNA vaccine: A vaccine targeting the hantavirus pulmonary syndrome (HPS) causative agent Andes Virus (ANDV), with potential pan-hantavirus effect. The plasmid backbone, pWRG7077, is modified to produce the active ingredient of the vaccine, plasmid pWRG/AND-M (opt2), and includes the ANDV M gene responsible for encoding viral GnGc envelope glycoproteins. ANDV DNA vaccine will be administered intramuscularly at 2 mg doses using the PharmaJet Stratis Needle-Free Injection System.
- 2 mg ANDV, 4 Dose Regimen: 2 mg (2 injections of 0.5 mL (1 mg/0.5 mL each)) of ANDV DNA vaccine intramuscularly into the left and right deltoid on Days 1, 29, 57 and 169 in a double-blinded manner. Sentinel subjects received all doses in an open label manner.
  Andes virus DNA vaccine: A vaccine targeting the hantavirus pulmonary syndrome (HPS) causative agent Andes Virus (ANDV), with potential pan-hantavirus effect. The plasmid backbone, pWRG7077, is modified to produce the active ingredient of the vaccine, plasmid pWRG/AND-M (opt2), and includes the ANDV M gene responsible for encoding viral GnGc envelope glycoproteins. ANDV DNA vaccine will be administered intramuscularly at 2 mg doses using the PharmaJet Stratis Needle-Free Injection System.
- 4 mg ANDV, 3 Dose Regimen: 4 mg (2 injections of 0.5 mL (2 mg/0.5 mL each)) of ANDV DNA vaccine intramuscularly into the left and right deltoid on Days 1, 29, 169 in a double-blinded manner. Sentinel subjects received all doses in an open label manner.
  Andes virus DNA vaccine: A vaccine targeting the hantavirus pulmonary syndrome (HPS) causative agent Andes Virus (ANDV), with potential pan-hantavirus effect. The plasmid backbone, pWRG7077, is modified to produce the active ingredient of the vaccine, plasmid pWRG/AND-M (opt2), and includes the ANDV M gene responsible for encoding viral GnGc envelope glycoproteins. ANDV DNA vaccine will be administered intramuscularly at 4 mg doses using the PharmaJet Stratis Needle-Free Injection System.
- 4 mg ANDV, 4 Dose Regimen: 4 mg (2 injections of 0.5 mL (2 mg/0.5 mL each)) of ANDV DNA vaccine intramuscularly into the left and right deltoid on Days 1, 29, 57 and 169 in a double-blinded manner. Sentinel subjects received all doses in an open label manner.
  Andes virus DNA vaccine: A vaccine targeting the hantavirus pulmonary syndrome (HPS) causative agent Andes Virus (ANDV), with potential pan-hantavirus effect. The plasmid backbone, pWRG7077, is modified to produce the active ingredient of the vaccine, plasmid pWRG/AND-M (opt2), and includes the ANDV M gene responsible for encoding viral GnGc envelope glycoproteins. ANDV DNA vaccine will be administered intramuscularly at 4 mg doses using the PharmaJet Stratis Needle-Free Injection System.
- Placebo: 2 mg (2 injections of 0.5 mL (1 mg/0.5 mL each)) or 4 mg (2 injections of 0.5 ml (2 mg/0.5 ml each)) of placebo intramuscularly into the left and right deltoid on Days 1, 29, 57, and 169 in a double-blinded manner.
  Placebo: Normal saline injections will be administered intramuscularly as matching placebo using the PharmaJet Stratis Needle-Free Injection System
Period: Overall Study
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo
Started | 10 | 10 | 10 | 10 | 8
Completed | 10 | 9 | 10 | 10 | 8
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: 2 mg (2 injections of 0.5 ml (1 mg/0.5 ml each)) or 4 mg (2 injections of 0.5 ml (2 mg/0.5 ml each)) of ANDV DNA vaccine intramuscularly into the left and right deltoid on Days 1, 29, 57, and 169 in a double-blinded manner.
  Placebo: Normal saline injections will be administered intramuscularly as matching placebo using the PharmaJet Stratis Needle-Free Injection System
- Total: Total of all reporting groups
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (6.8) | 33.8 (8.1) | 34.9 (8.9) | 35.9 (10.4) | 30.6 (8.8) | 34.7 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 9 | 7 | 4 | 33
  Male | 4 | 3 | 1 | 3 | 4 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 10 | 10 | 10 | 8 | 8 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 4 | 2 | 8
  White | 8 | 10 | 8 | 6 | 5 | 37
  More than one race | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Clinical Safety Laboratory Adverse Events
Description: Laboratory parameters include alanine aminotransferase (ALT), total bilirubin, creatinine, blood urea nitrogen (BUN), hemoglobin, absolute neutrophil count (ANC), sodium, potassium, white blood cells (WBC), and platelet count.
  Laboratory results were considered adverse events using the following thresholds: ALT 50 IU/L or greater; total bilirubin 1.30 mg/dL or greater; creatinine 0.81 mg/dL or greater (female) or 1.11 mg/dL or greater (male); BUN 24 mg/dL or greater; hemoglobin 11.6 g/dL or lower (female) or 13.2 g/dL or lower (male); ANC <1.8 K/mcL; sodium 135 mmol/L or lower (decrease) or 146 mmol/L or greater (increase); potassium 3.0 mmol/L or lower (decrease) or 5.2 mmol/L or greater (increase); WBC 4.4 K/mcL or lower (decrease) or 13.1 K/mcL or greater (increase 18 to <21 years) and 11.1 K/mcL or greater (increase 21 years or older); or platelets 134 K/mcL or below (decrease) or 467 K/mcL or greater (increase).
Time Frame: Day 8, Day 36, Day 64, Day 176
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Number; unit: participants
Groups:
- 2 mg ANDV, 3 Dose Regimen: 2 mg (2 injections of 0.5 mL (1 mg/0.5 mL each)) of ANDV DNA vaccine intramuscularly into the left and right deltoid on Days 1, 29, and 169 in a double-blinded manner. Sentinel subjects received all doses in an open label manner.
- 2 mg ANDV, 4 Dose Regimen: 2 mg (2 injections of 0.5 mL (1 mg/0.5 mL each)) of ANDV DNA vaccine intramuscularly into the left and right deltoid on Days 1, 29, 57 and 169 in a double-blinded manner. Sentinel subjects received all doses in an open label manner.
- 4 mg ANDV, 3 Dose Regimen: 4 mg (2 injections of 0.5 mL (2 mg/0.5 mL each)) of ANDV DNA vaccine intramuscularly into the left and right deltoid on Days 1, 29, 169 in a double-blinded manner. Sentinel subjects received all doses in an open label manner.
- 4 mg ANDV, 4 Dose Regimen: 4 mg (2 injections of 0.5 mL (2 mg/0.5 mL each)) of ANDV DNA vaccine intramuscularly into the left and right deltoid on Days 1, 29, 57 and 169 in a double-blinded manner. Sentinel subjects received all doses in an open label manner.
- Placebo: 2 mg (2 injections of 0.5 mL (1 mg/0.5 mL each)) or 4 mg (2 injections of 0.5 mL (2 mg/0.5 mL each)) of placebo intramuscularly into the left and right deltoid on Days 1, 29, 57, and 169 in a double-blinded manner.
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8
participants
  ALT : Day 36: number analyzed (Participants) | 9 | 10 | 10 | 10 | 7
  ALT : Day 36 | 0 | 2 | 0 | 0 | 0
  ALT : Day 64: number analyzed (Participants) | 9 | 10 | 10 | 10 | 7
  ALT : Day 64 | 0 | 2 | 0 | 0 | 0
  ALT : Day 176: number analyzed (Participants) | 9 | 9 | 10 | 9 | 5
  ALT : Day 176 | 2 | 0 | 0 | 0 | 0
  Total bilirubin : Day 8 | 0 | 0 | 0 | 0 | 1
  Total bilirubin : Day 36: number analyzed (Participants) | 9 | 10 | 10 | 10 | 7
  Total bilirubin : Day 36 | 1 | 0 | 0 | 0 | 0
  Total bilirubin : Day 64: number analyzed (Participants) | 9 | 10 | 10 | 10 | 7
  Total bilirubin : Day 64 | 0 | 0 | 1 | 0 | 0
  Total bilirubin : Day 176: number analyzed (Participants) | 9 | 9 | 10 | 9 | 5
  Total bilirubin : Day 176 | 0 | 0 | 1 | 0 | 0
  Creatinine : Day 8 | 0 | 1 | 2 | 5 | 0
  Creatinine : Day 36: number analyzed (Participants) | 9 | 10 | 10 | 10 | 7
  Creatinine : Day 36 | 1 | 1 | 2 | 4 | 0
  Creatinine : Day 64: number analyzed (Participants) | 9 | 10 | 10 | 10 | 7
  Creatinine : Day 64 | 0 | 0 | 1 | 4 | 0
  Creatinine : Day 176: number analyzed (Participants) | 9 | 9 | 10 | 10 | 5
  Creatinine : Day 176 | 1 | 0 | 3 | 3 | 0
  BUN : Day 8: number analyzed (Participants) | 0 | 1 | 2 | 4 | 0
  BUN : Day 8 |  | 1 | 2 | 4 |
  BUN : Day 36: number analyzed (Participants) | 0 | 1 | 2 | 4 | 0
  BUN : Day 36 |  | 1 | 2 | 4 |
  BUN : Day 64: number analyzed (Participants) | 0 | 0 | 1 | 4 | 0
  BUN : Day 64 |  |  | 1 | 4 |
  BUN : Day 176: number analyzed (Participants) | 1 | 0 | 3 | 3 | 0
  BUN : Day 176 | 1 |  | 3 | 3 |
  Hemoglobin : Day 8 | 0 | 1 | 0 | 1 | 0
  Hemoglobin : Day 36: number analyzed (Participants) | 9 | 10 | 10 | 10 | 7
  Hemoglobin : Day 36 | 1 | 1 | 1 | 1 | 0
  Hemoglobin : Day 64: number analyzed (Participants) | 9 | 10 | 10 | 10 | 7
  Hemoglobin : Day 64 | 1 | 1 | 1 | 1 | 1
  Hemoglobin : Day 176: number analyzed (Participants) | 9 | 9 | 10 | 9 | 5
  Hemoglobin : Day 176 | 2 | 1 | 0 | 1 | 0
  ANC : Day 8 | 0 | 0 | 1 | 0 | 0
  ANC : Day 36: number analyzed (Participants) | 9 | 10 | 10 | 10 | 7
  ANC : Day 36 | 0 | 0 | 1 | 0 | 0
  ANC : Day 64: number analyzed (Participants) | 9 | 10 | 10 | 10 | 7
  ANC : Day 64 | 0 | 2 | 0 | 1 | 0
  ANC : Day 176: number analyzed (Participants) | 9 | 9 | 10 | 9 | 5
  ANC : Day 176 | 0 | 1 | 0 | 1 | 0
  Sodium increase : Day 8 | 0 | 0 | 0 | 1 | 0
  Sodium increase : Day 36: number analyzed (Participants) | 9 | 10 | 10 | 10 | 7
  Sodium increase : Day 36 | 0 | 0 | 0 | 1 | 0
  WBC decrease : Day 8 | 0 | 1 | 1 | 0 | 0
  WBC decrease : Day 36: number analyzed (Participants) | 9 | 10 | 10 | 10 | 7
  WBC decrease : Day 36 | 0 | 2 | 1 | 0 | 0
  WBC decrease : Day 64: number analyzed (Participants) | 9 | 10 | 10 | 10 | 7
  WBC decrease : Day 64 | 0 | 3 | 1 | 1 | 0
  WBC decrease : Day 176: number analyzed (Participants) | 9 | 9 | 10 | 9 | 8
  WBC decrease : Day 176 | 0 | 2 | 1 | 1 | 0
  WBC increase : Day 8 | 1 | 0 | 1 | 0 | 0
  WBC increase : Day 36: number analyzed (Participants) | 9 | 10 | 10 | 10 | 7
  WBC increase : Day 36 | 1 | 0 | 0 | 1 | 0
  Platelets increased : Day 8 | 0 | 0 | 0 | 0 | 1
  Platelets increased : Day 64 | 0 | 1 | 0 | 1 | 0

2. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs) From Day 1 Through Day 337
Description: An adverse event was considered serious if it resulted in any of the following outcomes: death, a life-threatening adverse event (its occurrence places the participant at immediate risk of death), inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. Adverse events can be considered serious when they may jeopardize the patient or participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Day 1 through Day 337
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8
Participants | 0 | 0 | 0 | 1 | 0

3. Primary Outcome: Number of Participants Reporting Vaccine-Related Serious Adverse Events (SAEs) From Day 1 Through Day 337
Description: An adverse event is considered serious if it results in any of the following outcomes: death, a life-threatening adverse event (its occurrence places the participant at immediate risk of death), inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. Adverse events can be considered serious when they may jeopardize the patient or participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
  An adverse event was considered related to the study product if there was a reasonable possibility that the study product caused the adverse event. Reasonable possibility means that there is evidence to suggest a causal relationship between the study product and the adverse event.
Time Frame: Day 1 through Day 337
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8
Participants | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Experiencing Unsolicited Non-Serious Adverse Events at Any Time From Day 1 to Day 197
Description: Adverse events were defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. Unsolicited non-serious AEs were documented and reported from the time of first study vaccination through 28 days after the last study vaccination or after Day 169 if the fourth vaccination wasn't received.
Time Frame: Day 1 through Day 197
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8
Participants
  No unsolicited AEs | 4 | 2 | 1 | 2 | 3
  At least one unsolicited AE | 6 | 8 | 9 | 8 | 5

5. Primary Outcome: Number of Participants Experiencing Vaccine-Related Unsolicited Non-Serious Adverse Events at Any Time From Day 1 to Day 197
Description: Adverse events were defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. Unsolicited non-serious AEs were documented and reported from the time of first study vaccination through 28 days after the last study vaccination or after Day 169 if the fourth vaccination wasn't received.
  An adverse event was considered related to the study product if there was a reasonable possibility that the study product caused the adverse event. Reasonable possibility means that there is evidence to suggest a causal relationship between the study product and the adverse event.
Time Frame: Day 1 through Day 197
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8
Participants
  None | 8 | 8 | 8 | 7 | 6
  At least one related unsolicited AE | 2 | 2 | 2 | 3 | 2

6. Primary Outcome: Number of Participants Reporting Solicited Local Adverse Events From Day 1 Through Day 8
Description: Local adverse events solicited on a memory aid provided to participants included pain, tenderness, erythema, erythema measurement (measuring >0mm), induration, induration measurement (measuring >0mm), skin discoloration, ecchymosis, and ecchymosis measurement (measuring >0mm). Participants were considered to have experienced the AE if they reported an event of mild or greater severity on any of the 7 days following the first vaccination.
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Number; unit: participants
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8
participants
  Pain | 2 | 8 | 7 | 6 | 1
  Tenderness | 7 | 9 | 6 | 7 | 2
  Erythema | 7 | 9 | 8 | 4 | 3
  Erythema (measurement) | 7 | 9 | 8 | 4 | 3
  Induration | 4 | 10 | 7 | 7 | 3
  Induration (measurement) | 4 | 10 | 7 | 7 | 3
  Skin Discoloration | 2 | 2 | 2 | 2 | 0
  Ecchymosis | 2 | 4 | 3 | 3 | 2
  Ecchymosis (measurement) | 2 | 4 | 4 | 3 | 2

7. Primary Outcome: Number of Participants Reporting Solicited Local Adverse Events From Day 29 Through Day 36
Description: Local adverse events solicited on a memory aid provided to participants included pain, tenderness, erythema, erythema measurement (measuring >0mm), induration, induration measurement (measuring >0mm), skin discoloration, ecchymosis, and ecchymosis measurement (measuring >0mm). Participants were considered to have experienced the AE if they reported an event of mild or greater severity on any of the 7 days following the second vaccination.
Time Frame: Day 29 through Day 36
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Number; unit: participants
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8
participants
  Pain | 0 | 4 | 7 | 4 | 1
  Tenderness | 3 | 9 | 8 | 7 | 2
  Erythema | 7 | 9 | 8 | 5 | 3
  Erythema (measurement) | 7 | 9 | 8 | 6 | 3
  Induration | 4 | 10 | 6 | 7 | 3
  Induration (measurement) | 4 | 10 | 6 | 7 | 3
  Skin discoloration | 0 | 2 | 0 | 2 | 0
  Ecchymosis | 1 | 3 | 5 | 2 | 0
  Ecchymosis (measurement) | 1 | 3 | 6 | 2 | 0

8. Primary Outcome: Number of Participants Reporting Solicited Local Adverse Events From Day 57 Through Day 64
Description: Local adverse events solicited on a memory aid provided to participants included pain, tenderness, erythema, erythema measurement (measuring >0mm), induration, induration measurement (measuring >0mm), skin discoloration, ecchymosis, and ecchymosis measurement (measuring >0mm). Participants were considered to have experienced the AE if they reported an event of mild or greater severity on any of the 7 days following the third vaccination.
Time Frame: Day 57 through Day 64
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8
Participants
  Pain | 2 | 5 | 1 | 2 | 0
  Tenderness | 4 | 7 | 7 | 5 | 1
  Erythema | 7 | 10 | 6 | 6 | 2
  Erythema (Measurement) | 7 | 10 | 6 | 6 | 2
  Induration | 5 | 8 | 5 | 6 | 3
  Induration (Measurement) | 5 | 8 | 5 | 6 | 3
  Skin Discoloration | 0 | 0 | 1 | 2 | 0
  Ecchymosis | 1 | 5 | 1 | 3 | 0
  Ecchymosis (Measurement) | 1 | 5 | 1 | 3 | 0

9. Primary Outcome: Number of Participants Reporting Solicited Local Adverse Events From Day 169 Through Day 176
Description: Local adverse events solicited on a memory aid provided to participants included pain, tenderness, erythema, erythema measurement, induration, induration measurement, skin discoloration, ecchymosis, and ecchymosis measurement. Participants were considered to have experienced the AE if they reported an event of mild or greater severity on any of the 7 days following the fourth vaccination.
Time Frame: Day 169 through Day 176
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8
Participants
  Pain | 2 | 8 | 2 | 4 | 1
  Tenderness | 6 | 9 | 8 | 5 | 1
  Erythema | 7 | 9 | 10 | 6 | 2
  Erythema (Measurement) | 7 | 9 | 10 | 6 | 2
  Induration | 7 | 8 | 7 | 7 | 0
  Induration (Measurement) | 7 | 8 | 7 | 7 | 0
  Skin Discoloration | 2 | 3 | 1 | 1 | 0
  Ecchymosis | 3 | 3 | 2 | 3 | 0
  Ecchymosis (Measurement) | 3 | 3 | 2 | 3 | 0

10. Primary Outcome: Number of Participants Reporting Solicited Systemic Adverse Events From Day 1 Through Day 8
Description: Systemic adverse events solicited on a memory aid provided to participants included feverishness, malaise, fatigue, myalgia, headache, nausea, dizziness, and fever. Participants were considered to have experienced the AE if they reported an event of mild or greater severity on any of the 7 days following the first vaccination.
Time Frame: Day 1 through Day 8
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Number; unit: participants
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8
participants
  Feverishness | 0 | 0 | 1 | 1 | 0
  Malaise | 2 | 2 | 3 | 1 | 0
  Fatigue | 3 | 3 | 4 | 2 | 1
  Myalgia | 0 | 0 | 1 | 1 | 0
  Headache | 3 | 4 | 4 | 5 | 2
  Nausea | 0 | 1 | 1 | 1 | 1
  Diziness | 0 | 0 | 0 | 0 | 0
  Fever | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Participants Reporting Solicited Systemic Adverse Events From Day 29 Through Day 36
Description: Systemic adverse events solicited on a memory aid provided to participants included feverishness, malaise, fatigue, myalgia, headache, nausea, dizziness, and fever. Participants were considered to have experienced the AE if they reported an event of mild or greater severity on any of the 7 days following the second vaccination.
Time Frame: Day 29 through Day 36
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Number; unit: participants
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8
participants
  Feverishness | 0 | 0 | 1 | 1 | 0
  Malaise | 0 | 1 | 2 | 2 | 0
  Fatigue | 0 | 5 | 3 | 2 | 0
  Myalgia | 1 | 1 | 1 | 0 | 0
  Headache | 0 | 1 | 2 | 3 | 0
  Nausea | 0 | 0 | 0 | 0 | 0
  Dizziness | 0 | 0 | 2 | 0 | 0
  Fever | 0 | 0 | 0 | 1 | 0

12. Primary Outcome: Number of Participants Reporting Solicited Systemic Adverse Events From Day 57 Through Day 64
Description: Systemic adverse events solicited on a memory aid provided to participants included feverishness, malaise, fatigue, myalgia, headache, nausea, dizziness, and fever. Participants were considered to have experienced the AE if they reported an event of mild or greater severity on any of the 7 days following the third vaccination.
Time Frame: Day 57 through Day 64
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8
Participants
  Feverishness | 0 | 1 | 1 | 1 | 1
  Malaise | 0 | 3 | 2 | 1 | 1
  Fatigue | 1 | 5 | 2 | 2 | 1
  Myalgia | 0 | 2 | 1 | 1 | 0
  Headache | 2 | 4 | 2 | 2 | 0
  Nausea | 0 | 2 | 0 | 0 | 1
  Dizziness | 0 | 3 | 0 | 0 | 0
  Fever | 1 | 0 | 0 | 2 | 0

13. Primary Outcome: Number of Participants Reporting Solicited Systemic Adverse Events From Day 169 Through Day 176
Description: Systemic adverse events solicited on a memory aid provided to participants included feverishness, malaise, fatigue, myalgia, headache, nausea, dizziness, and fever. Participants were considered to have experienced the AE if they reported an event of mild or greater severity on any of the 7 days following the fourth vaccination.
  Systemic AEs were considered mild severity if they were noticeable but did not interfere with daily activity; events (other than headache) were considered moderate severity if they interfered with daily activity; events (other than headache) were considered severe severity if they caused significant interference and prevented daily activity. Headache events were considered moderate severity if they required any use of pain reliever or interfered with daily activity; headache events were severe if they prevented daily activity or required use of a prescription medication.
Time Frame: Day 169 through Day 176
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8
Participants
  Feverishness | 2 | 2 | 0 | 0 | 0
  Malaise | 3 | 1 | 1 | 2 | 0
  Fatigue | 3 | 4 | 1 | 1 | 0
  Myalgia | 2 | 1 | 1 | 0 | 0
  Headache | 3 | 2 | 1 | 3 | 1
  Nausea | 0 | 2 | 1 | 2 | 0
  Dizziness | 0 | 0 | 1 | 2 | 0
  Fever | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies to ANDV Measured by Plaque Reduction Neutralization Titers
Description: Venous blood was collected to perform a 50% plaque reduction neutralization test (PRNT) which was conducted with Andes Virus as the antigen. The geometric mean titer was calculated for each study arm from the results available at Day 1 prior to the first study vaccination, 28 days following the second study vaccination (and immediately prior to the third study vaccination; Day 57), 28 days following the third study vaccination (Day 85), and 28 days following the fourth study vaccination (Day 197).
  Results lower than the limit of detection (<20) were reported and analyzed as 14.1 (which is 20/ sqrt(2)).
Time Frame: Day 1, Day 57, Day 85, Day 197
Population: All participants in the intent-to-treat (ITT) population with valid results available at the given time point were included. Participants were included in the ITT population if they received at least one dose of study vaccine and contributed both pre- and at least one post-study vaccination for immunogenicity testing for which valid results (results are not missing and the laboratory did not deem the sample or results unfit for analysis) were reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8
titer
  Day 1 | 14.1 [NA to NA] — A confidence interval was not able to be computed for any arm at Day 1 due to a lack of variation in the data. | 14.1 [NA to NA] — A confidence interval was not able to be computed for any arm at Day 1 due to a lack of variation in the data. | 14.1 [NA to NA] — A confidence interval was not able to be computed for any arm at Day 1 due to a lack of variation in the data. | 14.1 [NA to NA] — A confidence interval was not able to be computed for any arm at Day 1 due to a lack of variation in the data. | 14.1 [NA to NA] — A confidence interval was not able to be computed for any arm at Day 1 due to a lack of variation in the data.
  Day 57: number analyzed (Participants) | 9 | 10 | 10 | 10 | 7
  Day 57 | 14.1 [11.4 to 27.7] | 24.6 [13.1 to 46.3] | 37.3 [13.9 to 99.7] | 24.6 [10.5 to 57.2] | 14.1 [NA to NA] — A confidence interval was not able to be computed due to a lack of variation in the data.
  Day 85 | 14.1 [NA to NA] — A confidence interval was not able to be computed due to a lack of variation in the data. | 45.9 [14.5 to 145.3] | 28.2 [13.1 to 60.8] | 34.8 [13.5 to 89.4] | 14.1 [NA to NA] — A confidence interval was not able to be computed due to a lack of variation in the data.
  Day 197: number analyzed (Participants) | 9 | 9 | 9 | 9 | 5
  Day 197 | 32.9 [11.8 to 91.8] | 68.5 [14.5 to 324.2] | 50.4 [17.6 to 143.9] | 217.7 [71.7 to 660.9] | 14.1 [NA to NA] — A confidence interval was not able to be computed due to a lack of variation in the data.

15. Secondary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies to ANDV Measured by Pseudovirion Neutralization Titers
Description: Venous blood was collected to perform a 50% pseudovirion neutralization assay (PsVNA) which was conducted with Andes Virus as the antigen. The geometric mean titer was calculated for each study arm from the results available at Day 1 prior to the first study vaccination, 28 days following the second study vaccination (and immediately prior to the third study vaccination; Day 57), 28 days following the third study vaccination (Day 85), and 28 days following the fourth study vaccination (Day 197).
  Results lower than the limit of detection (<20) were reported and analyzed as 14.1 (which is 20/ sqrt(2)).
Time Frame: Day 1, Day 57, Day 85, Day 197
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8
titer
  Day 1 | 14.1 [NA to NA] — A confidence interval was not able to be computed due to a lack of variation in the data. | 14.1 [12.9 to 17.6] | 14.1 [11.0 to 26.8] | 14.1 [NA to NA] — A confidence interval was not able to be computed due to a lack of variation in the data. | 14.1 [NA to NA] — A confidence interval was not able to be computed due to a lack of variation in the data.
  Day 57: number analyzed (Participants) | 9 | 10 | 10 | 10 | 7
  Day 57 | 22 [10.1 to 48] | 35.6 [15.8 to 80.4] | 200.1 [30.5 to 1312.4] | 68.8 [17.2 to 276.1] | 14.1 [NA to NA] — NA Explanation: A confidence interval was not able to be computed due to a lack of variation in the data.
  Day 85 | 14.1 [10.8 to 28.1] | 67.1 [19.3 to 233.6] | 119.4 [27.2 to 524.2] | 186.1 [38.2 to 905.9] | 14.1 [NA to NA] — NA Explanation: A confidence interval was not able to be computed due to a lack of variation in the data.
  Day 197: number analyzed (Participants) | 9 | 9 | 9 | 9 | 5
  Day 197 | 112.5 [16 to 791.8] | 230.5 [70.8 to 750.8] | 234.8 [50 to 1103.3] | 808.2 [168.2 to 3882.4] | 14.1 [NA to NA] — NA Explanation: A confidence interval was not able to be computed due to a lack of variation in the data.

16. Secondary Outcome: Number of Participants With ANDV Antibody Titers Greater Than or Equal to 20 as Measured by Plaque Reduction Neutralization Titers
Description: Venous blood was collected to perform a 50% plaque reduction neutralization test (PRNT) which was conducted with Andes Virus as the antigen. The number of participants with a titer greater than or equal to 20 was recorded for each study arm from the results available at 28 days following the second study vaccination (and immediately prior to the third study vaccination; Day 57), 28 days following the third study vaccination (Day 85), and 28 days following the fourth study vaccination (Day 197).
Time Frame: Day 57, Day 85, Day 197
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8
participants
  Day 57 | 2 | 4 | 4 | 2 | 0
  Day 85 | 0 | 4 | 4 | 4 | 0
  Day 197 | 4 | 4 | 6 | 8 | 0

17. Secondary Outcome: Number of Participants With ANDV Antibody Titers Greater Than or Equal to 20 as Measured by Pseudovirion Neutralization Titers
Description: Venous blood was collected to perform a 50% pseudovirion neutralization assay (PsVNA) which was conducted with Andes Virus as the antigen. The number of participants with a titer greater than or equal to 20 was recorded for each study arm from the results available at 28 days following the second study vaccination (and immediately prior to the third study vaccination; Day 57), 28 days following the third study vaccination (Day 85), 28 days following the fourth study vaccination (Day 197).
Time Frame: Day 57, Day 85, Day 197
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8
participants
  Day 57 | 2 | 5 | 6 | 5 | 0
  Day 85 | 1 | 5 | 6 | 7 | 0
  Day 197 | 5 | 9 | 8 | 8 | 0

18. Secondary Outcome: Percentage of Participants Achieving ANDV Antibody Seroconversion as Measured by Plaque Reduction Neutralization Titers
Description: Venous blood was collected to perform a 50% plaque reduction neutralization test (PRNT) which was conducted with Andes Virus as the antigen. A participant was considered to have seroconverted if their titer measured at least 40 if the baseline titer was less than 20, or if there was at least a 4-fold rise in titers from baseline if the baseline titer was greater than or equal to 20. The number of participants seroconverting was recorded for each study arm from the results at 28 days following the second study vaccination (and immediately prior to the third study vaccination; Day 57), 28 days following the third study vaccination (Day 85), and 28 days following the fourth study vaccination (Day 197).
Time Frame: Day 57, Day 85, Day 197
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8
percentage of participants
  Day 57 | 11.1 [0.3 to 48.2] | 30 [6.7 to 65.2] | 40 [12.2 to 73.8] | 20 [2.5 to 55.6] | 0 [0 to 41.0]
  Day 85 | 0 [0 to 30.8] | 40 [12.2 to 73.8] | 30 [6.7 to 65.2] | 40 [12.2 to 73.8] | 0 [0 to 36.9]
  Day 197: number analyzed (Participants) | 9 | 9 | 9 | 9 | 5
  Day 197 | 33.3 [7.5 to 70.1] | 44.4 [13.7 to 78.8] | 55.6 [21.2 to 86.3] | 88.9 [51.8 to 99.7] | 0 [0 to 36.9]

19. Secondary Outcome: Percentage of Participants Achieving ANDV Antibody Seroconversion at Day 57 as Measured by Pseudovirion Neutralization Titers
Description: Venous blood was collected to perform a 50% pseudovirion neutralization assay (PsVNA) which was conducted with Andes Virus as the antigen. A participant was considered to have seroconverted if their titer measured at least 40 if the baseline titer was less than 20, or if there was at least a 4-fold rise in titers from baseline if the baseline titer was greater than or equal to 20. The number of participants seroconverting was recorded for each study arm from the results at 28 days following the second study vaccination (and immediately prior to the third study vaccination; Day 57), 28 days following the third study vaccination (Day 85), and 28 days following the fourth study vaccination (Day 197).
Time Frame: Day 57, Day 85, Day 197
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 8
percentage of participants
  Day 57: number analyzed (Participants) | 9 | 10 | 10 | 10 | 7
  Day 57 | 22.2 [2.8 to 60] | 30 [6.7 to 65.2] | 60 [26.2 to 87.8] | 50 [18.7 to 81.3] | 0 [0 to 41]
  Day 85 | 10 [0.3 to 44.5] | 40 [12.2 to 73.8] | 60 [26.2 to 87.8] | 70 [34.8 to 93.3] | 0 [0 to 36.9]
  Day 197: number analyzed (Participants) | 9 | 9 | 9 | 9 | 5
  Day 197 | 55.6 [21.2 to 86.3] | 77.8 [40 to 97.2] | 88.9 [51.8 to 99.7] | 88.9 [51.8 to 99.7] | 0 [0 to 52.2]

ADVERSE EVENTS:
Time Frame: Non-serious AEs were collected through 28 days following the final vaccination, up to Day 197; SAEs were collected through Day 337.
Arm/Group | 2 mg ANDV, 3 Dose Regimen | 2 mg ANDV, 4 Dose Regimen | 4 mg ANDV, 3 Dose Regimen | 4 mg ANDV, 4 Dose Regimen | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 1/10 | 0/8
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 10/10 | 10/10 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 mg ANDV, 3 Dose Regimen (N=10) | 2 mg ANDV, 4 Dose Regimen (N=10) | 4 mg ANDV, 3 Dose Regimen (N=10) | 4 mg ANDV, 4 Dose Regimen (N=10) | Placebo (N=8)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Acute Rhabdomyolysis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 mg ANDV, 3 Dose Regimen (N=10) | 2 mg ANDV, 4 Dose Regimen (N=10) | 4 mg ANDV, 3 Dose Regimen (N=10) | 4 mg ANDV, 4 Dose Regimen (N=10) | Placebo (N=8)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 5 (6) | 4 (4) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (5) | 2 (2) | 2 (3) | 2 (2)
Fatigue (General disorders) | 4 (7) | 7 (17) | 6 (10) | 4 (7) | 2 (2)
Feeling of body temperature change (General disorders) | 2 (2) | 3 (3) | 2 (3) | 3 (3) | 1 (1)
Injection site haemorrhage (General disorders) | 3 (7) | 6 (15) | 6 (12) | 4 (11) | 2 (2)
Malaise (General disorders) | 4 (5) | 5 (7) | 5 (8) | 3 (6) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Vaccination site discolouration (General disorders) | 3 (4) | 4 (7) | 2 (2) | 4 (7) | 0 (0)
Vaccination site erythema (General disorders) | 9 (28) | 10 (37) | 10 (32) | 8 (22) | 6 (10)
Vaccination site pain (General disorders) | 8 (20) | 10 (34) | 8 (30) | 9 (26) | 6 (9)
Vaccination site induration (General disorders) | 9 (20) | 10 (36) | 9 (25) | 10 (27) | 5 (9)
Blood bilirubin increased (Investigations) | 3 (3) | 0 (0) | 1 (7) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 2 (4) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (2) | 1 (3) | 3 (11) | 6 (25) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (11) | 1 (9) | 1 (2) | 1 (5) | 1 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (3) | 1 (5) | 2 (3) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 5 (10) | 1 (7) | 2 (3) | 1 (1)
White blood cell count increased (Investigations) | 2 (2) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 2 (4) | 1 (2) | 0 (0)
Diziness (Nervous system disorders) | 0 (0) | 3 (4) | 3 (3) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 5 (8) | 6 (11) | 7 (10) | 5 (14) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT03682107/Prot_001.pdf
  • Statistical Analysis Plan (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/07/NCT03682107/SAP_002.pdf
  • Informed Consent Form (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/07/NCT03682107/ICF_000.pdf